CLINICAL TRIAL: NCT00986856
Title: A Phase IV Study Comparing Clinical and Bacteriological Efficacy of Fucidin® Cream With Fucidin® Cream Vehicle in the Treatment of Impetigo in Paediatric Patients
Brief Title: Fucidin® Cream in the Treatment of Impetigo
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment failed
Sponsor: LEO Pharma (Industry)
Responsible Party: Pontus Hegardt, Clinical Trial Manager, LEO Pharma
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUC 0301 INT
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2015-03

CONDITIONS: Impetigo
MeSH Terms: conditions — Impetigo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fucidin® cream (Experimental)
  Interventions: Drug: Fucidin® cream
- Fucidin® cream vehicle (Placebo Comparator)
  Interventions: Drug: Fucidin® cream

INTERVENTIONS:
Drug: Fucidin® cream

SUMMARY:
To investigate the clinical and bacteriological efficacy of Fucidin® cream in the treatment of impetigo in paediatric patients.

To assess the validity of in vitro susceptibility-testing of S. aureus to fusidic acid as a prediction of clinical and bacteriological outcome in impetigo patients treated with Fucidin® cream.

To investigate the genetic relationship between S. aureus-strains isolated from impetigo patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of impetigo,
* Patients aged 2-11 years,
* Patients of either sex,
* Patients whose parent(s) has(ve) provided written consent, AND
* Patients with a severity score of 1 for at least one of the following signs: pustules/infected bullae, erythema and infiltration/induration.

Exclusion Criteria:

* Patients with other active inflammatory dermatitis at the area of impetigo,
* Patients with a temperature above 38.5 C rectally (or equivalent), OR
* Patients who have been administered topical or systemic Fucidin® or other antibacterial agents within the previous 4 weeks.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2004-05; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (2):
- Institute of Internal Medicin, Haukeland University Hospital, Bergen, Norway
- Vårdcentrum Kungshöjd, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Groups:
- Fucidin® Cream: Fucidin® cream 20 mg/g 3 times daily for 10 days
- Fucidin® Cream Vehicle: Fucidin® cream vehicle 3 times daily for 10 days
Period: Overall Study
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Started | 42 | 16
Completed | 42 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle | Total
Number analyzed (Participants) | 42 | 16 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 16 | 58
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.8 (2.7) | 6.3 (2.9) | 5.2 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 8 | 26
  Male | 24 | 8 | 32
Region of Enrollment [Number; unit: participants]
  Sweden | 32 | 15 | 47
  Norway | 10 | 1 | 11
S.aureus susceptible to fusidic acid [Number; unit: S. aureus]
  S. aureus susceptible to fusidic acid | 12 | 4 | 16
  S. aureus resistant to fusidic acid | 18 | 8 | 26
  No S. aureus isolated | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Success (Marked Improvement or Completely Cleared) and Bacteriological Success (Eradication) at End of Treatment (EOT).
Time Frame: EOT: Visit at Day 25
Population: The analysis population was the full (intention-to treat) analysis set including the patients with confirmed presence of pathogenic bacteria (S. aureus and/or betahaemolytic streptococci (group A)) at baseline
Measure: Number; unit: Participants
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Number analyzed (Participants) | 33 | 13
Participants
  Clinical and bacteriological success | 16 | 1
  Clinical and bacteriological failure | 17 | 12
Statistical Analysis 1: Comparison: Fucidin® Cream vs Fucidin® Cream Vehicle; Test type: Superiority or Other; p < 0.01, Cochran-Mantel-Haenszel — Test for the hypothesis of odds ratio equal to 1; Odds Ratio (OR) = 13.2, 95% CI [1.4 to 120.4]

2. Secondary Outcome: Number of Patients With Clinical Success at Visit 2
Time Frame: Visit 2: Day 4
Population: The full analysis set consists of 56 patients, 40 patients in the Fucidin® cream 20 mg/g group and 16 patients in the Fucidin® cream vehicle group (2 patients excluded because of lack of efficacy data)
Measure: Number; unit: Participants
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Number analyzed (Participants) | 40 | 16
Participants
  Success | 18 | 2
  Failure | 22 | 14
Statistical Analysis 1: Comparison: Fucidin® Cream vs Fucidin® Cream Vehicle; Test type: Superiority or Other; p = 0.023, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.7, 95% CI [1.1 to 28.6]

3. Secondary Outcome: Number of Patients With Clinical Success at Visit 3
Time Frame: Visit 3: Day 11
Population: The analysis population were those patients who had a visit 3 observation
Measure: Number; unit: Participants
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Number analyzed (Participants) | 34 | 10
Participants
  Success | 27 | 7
  Failure | 7 | 3
Statistical Analysis 1: Comparison: Fucidin® Cream vs Fucidin® Cream Vehicle; Test type: Superiority or Other; p = 0.54, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.3 to 8.1]

4. Secondary Outcome: Number of Patients With Clinical Success at EOT
Time Frame: EOT: Visit at day 25
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Number analyzed (Participants) | 40 | 16
Participants
  Success | 27 | 7
  Failure | 13 | 9
Statistical Analysis 1: Comparison: Fucidin® Cream vs Fucidin® Cream Vehicle; Test type: Superiority or Other; p = 0.1, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.7, 95% CI 2-sided [0.8 to 8.8]

5. Secondary Outcome: Number of Patients With Bacteriological Success at Visit 2
Time Frame: Visit 2: Day 4
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Number analyzed (Participants) | 33 | 13
Participants
  Success | 6 | 0
  Failure | 27 | 13
Statistical Analysis 1: Comparison: Fucidin® Cream vs Fucidin® Cream Vehicle; Test type: Superiority or Other; p = 0.1, Cochran-Mantel-Haenszel

6. Secondary Outcome: Number of Patients With Bacteriological Success at Visit 3
Time Frame: Visit 3: Day 11
Population: The analysis population were those patients who had a visit 3 observation
Measure: Number; unit: Participants
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Number analyzed (Participants) | 27 | 6
Participants
  Success | 17 | 1
  Failure | 10 | 5
Statistical Analysis 1: Comparison: Fucidin® Cream vs Fucidin® Cream Vehicle; Test type: Superiority or Other; p = 0.043, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.5, 95% CI [0.9 to 83.5]

7. Secondary Outcome: Number of Patients With Bacteriological Success at EOT
Time Frame: EOT: Visit at day 25
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Number analyzed (Participants) | 33 | 13
Participants
  Success | 17 | 1
  Failure | 16 | 12
Statistical Analysis 1: Comparison: Fucidin® Cream vs Fucidin® Cream Vehicle; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 12.8, 95% CI [1.5 to 109.6]

8. Secondary Outcome: The Actual Change in Total Severity Score From Baseline to End of Treatment (LOCF).
Description: Total Severity Score is the sum of scores for the following 5 signs: Pustules/infected bullae, erythema, infiltration/induration, erosions and crusting. Each sign is assessed using a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe involvement. Minimum Total Severity score is 0, maximum score is 15.
Time Frame: EOT: Visit at day 25
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Number analyzed (Participants) | 40 | 16
Units on a scale | -3.9 (3.5) | -1.2 (4.4)
Statistical Analysis 1: Comparison: Fucidin® Cream vs Fucidin® Cream Vehicle; Test type: Superiority or Other; p = 0.008, Regression, Linear; Mean Difference (Final Values) = -2.8, 95% CI [-4.8 to -0.8], Standard Deviation 2

ADVERSE EVENTS:
Description: All 58 randomised patients comprised the safety analysis set except patients who: 1. did not provide any post randomisation safety data or 2. did not use any trial medication confirmed by return of all trial medication given to the patients.
Arm/Group | Fucidin® Cream | Fucidin® Cream Vehicle
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/16
Other Adverse Events (participants affected / at risk) | 5/40 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fucidin® Cream (N=40) | Fucidin® Cream Vehicle (N=16)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 3 (3) | 4 (4)
Infections and (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
It was planned to Incl. 360 Pts(Proport.3:1 Fucidin® cream:Fucidin® cream vehicle), but due to very slow recruitment in SE and N and inability to Incl. UK, only 59 Pts were enrolled. 58 Pts were randomised: 42Fucidin® cream:16 Fucidin® cream vehicle.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No